CLINICAL TRIAL: NCT01042886
Title: Partnerships to Overcome Obesity Disparities in Hawaii
Brief Title: PILI 'Ohana Project: Partnerships to Overcome Obesity Disparities in Hawaii (3-Year Pilot)
Acronym: PILI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Marjorie K. Mau/Principal Investigator, Department of Native Hawaiian Health, University of Hawaii at Manoa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R24MD001660-03 (NIH); R24MD001660 (NIH)
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Overweight; Obesity
Keywords: Non-blind, randomized controlled trial; Pilot study
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family plus community focused intervention (Experimental)
  Interventions: Behavioral: PILI 'Ohana Lifestyle Program
- Standard Behavioral Weight Loss Maintenance Intervention (Active Comparator)
  Interventions: Behavioral: Standard Behavioral Weight Loss Maintenance Program

INTERVENTIONS:
Behavioral: PILI 'Ohana Lifestyle Program — 9-month weight loss and weight loss maintenance intervention focusing on family and community resources/supports.
  Arms: Family plus community focused intervention
Behavioral: Standard Behavioral Weight Loss Maintenance Program — 9-month weight loss and weight loss maintenance intervention based on empirically-supported behavioral foci and strategies.
  Arms: Standard Behavioral Weight Loss Maintenance Intervention

SUMMARY:
The PILI 'Ohana CBPR partnership implemented a pilot study to determine whether a Family plus Community focused intervention will improve weight loss maintenance compared to Standard follow-up in overweight/obese Native Hawaiian (NH) and other Pacific People (PP) adults (> 18 yr. old) after receiving a standard individual-focused behavioral intervention. The primary hypothesis was that overweight/obese NH and PP adults that undergo a combined family-focused plus community-focused intervention vs. a standard follow-up after receiving a standard individual-focused behavioral intervention will have significantly higher rates of weight loss maintenance.

DETAILED DESCRIPTION:
The long term mission of the PILI 'Ohana Program is to integrate community wisdom and expertise with scientific methods to conduct research on health disparities with a specific emphasis on obesity in NHs and PPs. Recognizing that recent advances in medicine such as the reduction of cardiovascular disease mortality and the prevention of type 2 diabetes mellitus, have not translated into benefits for all sectors of the U.S. population, especially ethnic and racial minority populations, the PILI 'Ohana Program aims to address this gap through community-academic partnerships focused on interventions to promote change in obesity-related disparities in NH and PP communities. One of the scientific goals of the PILI 'Ohana Program focused on designing and implementing research activities aimed at completing a pilot intervention study to provide the basis for a more definitive, hypothesis-driven 5-year research study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Native Hawaiian, Filipino or other Pacific Islander ethnic background;
* Age 18 years or older;
* Overweight or Obese defined as BMI > 25 kg/m2 (NH or Pacific Islanders) or > 23 kg/m2 (Filipino ethnic background);
* Willing and able to follow a behavioral weight loss intervention program that could potentially include 150 minutes of brisk walking per week (or equivalent) and a dietary regimen designed to induce weight loss of ~1-2 lbs per week;
* Able to identify at least 2-3 family, friends or co-workers that would be willing to support the participant during the course of the study.

Exclusion Criteria:

* Survival less than 6 months;
* Planning to move out of the community during the intervention study period (16 months);
* Pregnancy;
* Any dietary or exercise restrictions that would prevent an individual from fully participating in the intervention protocol (i.e. end stage renal disease on a renal diet, etc.);
* Any co-morbid condition (physical and mental disabilities) that would prevent the individual from participating in the intervention protocol (i.e. severe arthritis, hemi-paresis, major psychiatric illness, eating disorders, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Weight in kilograms (kg) | Baseline, 3-month follow-up, and 9-month follow-up
Physical functioning measured by a 6-minute walk test | Baseline, 3-month follow-up, and 9-month follow-up

SECONDARY OUTCOMES:
Blood pressure | Baseline, 3-month follow-up, and 9-month follow-up
Change in dietary fat intake based on self-report | Baseline, 3-month follow-up, and 9-month follow-up
Change in physical activity level based on self-report | Baseline, 3-month follow-up, and 9-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Kaholokula, PhD, Study Director — University of Hawaii at Manoa; Marjorie K Mau, MD, Principal Investigator — University of Hawaii at Manoa
Locations (1):
- Department of Native Hawaiian Health, University of Hawaii, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Kaholokula JK, Townsend CK, Ige A, Sinclair Ki, Mau MK, Leake A, Palakiko DM, Yoshimura SR, Kekauoha P, Hughes C. Sociodemographic, behavioral, and biological variables related to weight loss in native Hawaiians and other Pacific Islanders. Obesity (Silver Spring). 2013 Mar;21(3):E196-203. doi: 10.1002/oby.20038. PMID 23404724
- [Derived] Sinclair KA, Makahi EK, Shea-Solatorio C, Yoshimura SR, Townsend CK, Kaholokula JK. Outcomes from a diabetes self-management intervention for Native Hawaiians and Pacific People: Partners in Care. Ann Behav Med. 2013 Feb;45(1):24-32. doi: 10.1007/s12160-012-9422-1. PMID 23086589
- [Derived] Kaholokula JK, Mau MK, Efird JT, Leake A, West M, Palakiko DM, Yoshimura SR, Kekauoha BP, Rose C, Gomes H. A family and community focused lifestyle program prevents weight regain in Pacific Islanders: a pilot randomized controlled trial. Health Educ Behav. 2012 Aug;39(4):386-95. doi: 10.1177/1090198110394174. Epub 2011 May 6. PMID 21551421